CLINICAL TRIAL: NCT04221893
Title: Phase II Study of Hypofractionated Radiation Therapy to Augment Immune Response in Patients With Metastatic GastroIntestinal Malignancies Progressing on Immune Therapy (ARM-GI)
Brief Title: Radiation Therapy for the Treatment of Metastatic Gastrointestinal Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19721; NCI-2019-08355 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Stage IV Esophageal Adenocarcinoma; Stage IV Esophageal Squamous Cell Carcinoma; Stage IV Gastric Cancer; Stage IV Adenocarcinoma of the Gastroesophageal Junction; Stage IVA Esophageal Adenocarcinoma; Stage IVA Esophageal Squamous Cell Carcinoma; Stage IVA Gastric Cancer; Stage IVA Adenocarcinoma of the Gastroesophageal Junction; Stage IVB Esophageal Adenocarcinoma; Stage IVB Esophageal Squamous Cell Carcinoma; Stage IVB Gastric Cancer; Stage IVB Gastroesophageal Junction Adenocarcinoma; Metastatic Anal Canal Carcinoma; Metastatic Colorectal Carcinoma; Metastatic Esophageal Carcinoma; Metastatic Gastric Carcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Metastatic Hepatocellular Carcinoma; Metastatic Malignant Digestive System Neoplasm; Metastatic Small Intestinal Carcinoma; Pancreatobiliary Carcinoma; Pathologic Stage IV Gastric Cancer AJCC v8; Pathologic Stage IVA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IVA Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IVB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IVB Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IV Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IV Gastric Cancer AJCC v8; Postneoadjuvant Therapy Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVA Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVA Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVB Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVB Esophageal Squamous Cell Carcinoma AJCC V8; Postneoadjuvant Therapy Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Stage IV Anal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVA Hepatocellular Carcinoma AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVB Hepatocellular Carcinoma AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Stomach Neoplasms; Anal Canal Carcinoma; Colorectal Neoplasms; Esophageal Neoplasms; Carcinoma, Hepatocellular; Gastrointestinal Neoplasms; Anus Neoplasms | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Radiation therapy (RT) (Experimental): Patients undergo radiation therapy for a total of 5 treatments over 5-9 calendar days in the absence of disease progression or unacceptable toxicity. Target prescription dose will be 30 Gy in 5 fractions and each treatment site (up to 5) will undergo standard Department-approved treatment planning, quality-assurance, and delivery protocols
  Interventions: Radiation: Radiation Therapy (RT)

INTERVENTIONS:
Radiation: Radiation Therapy (RT) — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; irradiated; Irradiation; RADIATION; Radiation Therapy; Radiation Therapy, Not otherwise specified; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase II trial studies how well radiation therapy works for the treatment of gastrointestinal cancer that are spreading to other places in the body (metastatic). Radiation therapy uses high energy x-rays to kill cancer cells and shrink tumors. This trial is being done to determine if giving radiation therapy to patients who are being treated with immunotherapy and whose cancers are progressing (getting worse) can slow or stop the growth of their cancers. It may also help researchers determine if giving radiation therapy to one tumor can stimulate the immune system to attack other tumors in the body that are not targeted by the radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether radiation therapy can convert overall response rates from progressive disease to stable or responsive disease as measured by Response Evaluation Criteria in Solid Tumors (RECIST) version (v.) 1.1.

SECONDARY OBJECTIVES:

I. To define overall response rate by immune-Modified Response Evaluation Criteria in Solid Tumors (iRECIST) criteria.

II. To determine time to progression. III. To determine overall survival. IV. To determine local control in radiated lesion(s). V. To characterize the effect of distant radiation on unirradiated target lesions.

VI. To describe the incidence of new metastatic lesions. VII. To determine treatment safety by Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0.

VIII. To describe time to new systemic therapy.

EXPLORATORY OBJECTIVES:

I. To define radiation-induced effects on circulating immune cells. II. To describe remodeling of the circulating T cell repertoire by deep sequencing of variable, diversity and joining (VDJ) regions of T cell receptors (TCRs).

III. To describe changes in circulating tumor deoxyribonucleic acid (DNA) (ctDNA).

OUTLINE:

Patients undergo radiation therapy for a total of 5 treatments over 5-9 calendar days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 14 day, 6 months, and then up to 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically, cytologically, or radiographically confirmed metastatic gastrointestinal (GI) malignancy (esophageal, gastroesophageal, gastric, small intestine, hepatocellular, pancreaticobiliary, colorectal, or anal cancer).
2. Patients must be receiving immunotherapy (checkpoint inhibitor or CTLA4 inhibitor) with overall response of progressive disease by RECIST criteria.
3. Patients must have at least two metastases which are individually progressing as per RECIST criteria, one of which can be safely unirradiated as adjudicated by the treating radiation oncologist (e.g. lesions for which small increases in dimensions are unlikely to precipitate significant symptoms).
4. Patients must have 1-5 sites of disease meeting standard-of-care indications for palliative radiation therapy as adjudicated by the treating radiation oncologist. For example:

   * Symptomatic disease causing pain, bleeding, dyspnea, dysphagia, or nausea
   * At-risk for neurologic, respiratory, cardiovascular, gastrointestinal, musculoskeletal, or hepatobiliary compromise
5. Evaluation by a radiation oncologist within 28 days of study registration.
6. Must have adequate organ function to administer radiation therapy and immunotherapy as per standard of care.
7. Age >= 18 years.
8. Life expectancy exceeding 6 months.
9. Eastern Cooperative Oncology Group (ECOG) 0-2 or Karnofsky performance status >= 50.
10. Radiation therapy is known to be teratogenic and therefore women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of radiation therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for 3 months after completion of radiation therapy. Contraception requirements during the follow-up period of 6 months will be according to standard of care for immunotherapy administration.

    a. If a woman is of child-bearing potential, a negative pregnancy test within 28 days prior to study enrollment is required.
11. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Enrollment on immunotherapy clinical trial for which radiation therapy is not permitted.
2. Administration of radiation therapy within 4 weeks prior to study enrollment.
3. Treatment with systemic corticosteroids or other immunosuppressive medications which would significantly diminish the effect of immunotherapy as judged by the treating physician.
4. Radiation therapy is contraindicated as adjudicated by the radiation oncologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 8 weeks
  Proportion of patients who achieve as their best overall response according to Response Evaluation Criteria in Solid Tumors (RECIST) v. 1.1 criteria: Stable disease (SD), partial response (PR), confirmed Complete Response (CR), or progressive disease (PD). Corresponding exact confidence intervals will be reported for the entire cohort and stratified by histologic subtype, programmed cell death protein 1 (PD-1)/programmed death-ligand 1 (PD-L1) status, microsatellite instability (MSI), and organs treated if sample size allows. Patients with unevaluable or unknown response status will be considered nonresponders.

SECONDARY OUTCOMES:
ORR by immune-Modified Response Evaluation Criteria in Solid Tumors (iRECIST) | Up to 8 weeks
  Will be determined by immune-Modified Response Evaluation Criteria in Solid Tumors (iRECIST). Immune Complete Response (iCR), Partial Response (iPR), or Stable Disease (iSD) per definitions of CR, PR, and SD, but occurring after initial immune unconfirmed progressive disease (iUPD). The same definition will be used for per lesion analysis. PD will be designated for all patients with PD determination by RECIST v1.1 or immune-confirmed progressive disease (iCPD) by iRECIST. Unconfirmed response for all patients designated as iUPD. Will be reported as proportion of response and corresponding exact confidence intervals. Patients with unevaluable or unknown response status will be considered nonresponders.
Progression free survival (PFS) | Up to 36 months
  PFS is defined as the duration of time from start of radiation treatment to time of progression or death a proportion with exact confidence intervals and will be reported for the entire cohort and stratified by histologic subtype, PD1/PDL1 status, MSI, and organs treated if sample size allows. Time to local progression will be described using the cumulative incidence method and comparisons between strata via Gray's test, if sample size allows; Otherwise, Kaplan-Meier methodology will be used and comparisons will be made via log-rank test; and Cox proportional hazards analysis, if possible.
Overall survival (OS) | Up to 36 months
  OS will be measured from the date of initiation of RT. OS is defined as the time from the date of initiation of RT to the date of death due to any cause. Censoring will be performed using the date of last known contact for those who are alive at the time of analysis. OS will be reported for the entire cohort and stratified by histologic subtype, PD1/PDL1 status, MSI, and organs treated if sample size allows.
Determine local control in radiated lesion(s) | Up to 36 months
  Local control will be defined as absence of per-lesion PD in an irradiated lesion (as defined above, a 20% increase in the longest diameter since the treatment started or a 5 mm increase over the nadir longest diameter from initiation of radiation therapy to time of progression of radiated lesion(s)
Tumor measurement change by RECIST or iRECIST | Up to 8 weeks
  Abscopal response rate is defined as present for all patients for whom an unirradiated target or non-target lesion previously determined to be a progressing lesion is designated as SD, CR/iCR or PR/iPR on per-lesion analysis will be described as a proportion with exact confidence intervals and will be reported for the entire cohort, reported for RECIST and iRECIST definitions, and stratified by histologic subtype, PD1/PDL1 status, MSI, and organs treated if sample size allows
Incidence of New metastatic lesions | Up to 8 weeks
  From initiation of radiation therapy to first imaging scan after radiation therapy completion, time to new metastatic lesions will be described using the cumulative incidence method and comparisons between strata via Gray's test, if sample size allows; Kaplan-Meier methodology will be used and comparisons will be made via log-rank test; and Cox proportional hazards analysis, if possible.
Frequency of grade 3 or higher adverse events | Up to 36 months
  Common Terminology Criteria for Adverse Events (CTCAE v.5.0) will be used to determine frequency of grade 3 or higher adverse events reported as a proportion with corresponding exact confidence intervals.
Time to new systemic therapy | Up to 36 months
  Time to new systemic therapy from initiation of radiation therapy to initiation of new systemic therapy will be described using Kaplan-Meier product limit estimators, and Cox proportional hazards analysis, if possible.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Feng, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California

IPD SHARING:
Plan to Share IPD: No